CLINICAL TRIAL: NCT02578680
Title: A Randomized, Double-Blind, Phase III Study of Platinum+Pemetrexed Chemotherapy With or Without Pembrolizumab (MK-3475) in First Line Metastatic Non-squamous Non-small Cell Lung Cancer Subjects (KEYNOTE-189)
Brief Title: Study of Pemetrexed+Platinum Chemotherapy With or Without Pembrolizumab (MK-3475) in Participants With First Line Metastatic Nonsquamous Non-small Cell Lung Cancer (MK-3475-189/KEYNOTE-189)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3475-189; 163421 (Registry Identifier: JAPIC-CTI); MK-3475-189 (Other: MSD); 2015-003694-15 (EudraCT Number)
Record Dates: First submitted 2015-10-15; First posted 2015-10-19 (Estimated); Results first posted 2018-11-28 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: PD1; PD-1; PDL1; PD-L1; Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Cisplatin; Carboplatin; Pemetrexed; Folic Acid; Vitamin B 12; Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) PLUS pemetrexed 500 mg/m^2 IV (with vitamin supplementation) PLUS cisplatin 75 mg/m^2 IV OR carboplatin Area Under the Curve (AUC) 5 IV on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by pembrolizumab 200 mg IV PLUS pemetrexed 500 mg/m^2 IV Q3W until progression. (Participants who receive pembrolizumab 200 mg IV Q3W for up to 2 years but experience disease progression, will be eligible to receive a second course of pembrolizumab monotherapy 200 mg IV Q3W, at the investigator's discretion, for up to 1 additional year.)
  Interventions: Biological: Pembrolizumab 200 mg; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Dietary Supplement: Folic acid 350-1000 μg; Dietary Supplement: Vitamin B12 1000 μg; Drug: Dexamethasone 4 mg
- Control (Active Comparator): Participants receive saline placebo IV PLUS pemetrexed 500 mg/m^2 IV (with vitamin supplementation) PLUS cisplatin 75 mg/m^2 IV OR carboplatin AUC 5 IV on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by saline placebo IV PLUS pemetrexed 500 mg/m^2 IV Q3W until progression. (Effective 23-Dec-2019, participants will discontinue saline placebo. If documented progression occurs, participants may be able to receive pembrolizumab monotherapy Q3W for the remainder of the study.)
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed; Dietary Supplement: Folic acid 350-1000 μg; Dietary Supplement: Vitamin B12 1000 μg; Drug: Dexamethasone 4 mg; Drug: Saline solution

INTERVENTIONS:
Biological: Pembrolizumab 200 mg — IV infusion
  Arms: Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed
Drug: Cisplatin — IV infusion
Drug: Carboplatin — IV infusion
Drug: Pemetrexed — IV infusion
Dietary Supplement: Folic acid 350-1000 μg — Orally; at least 5 doses of folic acid must be taken during the 7 days preceding the first dose of pemetrexed, and folic acid dosing must continue during the full course of therapy and for 21 days after the last dose of pemetrexed.
Dietary Supplement: Vitamin B12 1000 μg — Intramuscular injection in the week preceding the first dose of pemetrexed and once every 3 cycles thereafter. Subsequent vitamin B12 injections may be given the same day as pemetrexed administration.
Drug: Dexamethasone 4 mg — For prophylaxis; orally twice per day (or equivalent). Taken the day before, day of, and day after pemetrexed administration.
Drug: Saline solution — IV infusion
  Arms: Control

SUMMARY:
This is an efficacy and safety study of pembrolizumab (MK-3475) combined with pemetrexed/platinum chemotherapy versus pemetrexed/platinum chemotherapy alone in participants with advanced or metastatic nonsquamous non-small cell lung cancer (NSCLC) who have not previously received systemic therapy for advanced disease. Participants will be randomly assigned to receive pembrolizumab combined with pemetrexed/platinum (Investigators choice of cisplatin or carboplatin), OR pemetrexed/platinum (Investigators choice of cisplatin or carboplatin).

With Amendment 10 (effective date 23-Dec-2019), active participants, investigator, and sponsor personnel or delegate(s) involved in the treatment administration or clinical evaluation of the participants will be unblinded, and all participants in the 'control' arm will discontinue saline placebo.

With Amendment 11 (effective date 31-Jan-2022), once the study objectives have been met or the study has ended, participants will be discontinued from this study and will be enrolled in an extension study to continue protocol-defined assessments and treatment.

The primary hypothesis is that pembrolizumab in combination with pemetrexed/platinum chemotherapy prolongs Progression-Free Survival (PFS) and Overall Survival (OS) compared to pemetrexed/platinum chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically-confirmed or cytologically confirmed diagnosis of stage IV nonsquamous NSCLC.
* Has confirmation that epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK)-directed therapy is not indicated.
* Has measurable disease.
* Has not received prior systemic treatment for their advanced/metastatic NSCLC.
* Can provide tumor tissue.
* Has a life expectancy of at least 3 months.
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status.
* Has adequate organ function
* If female of childbearing potential, is willing to use adequate contraception for the course of the study through 120 days after the last dose of study medication or through 180 days after last dose of chemotherapeutic agents.
* If male with a female partner(s) of child-bearing potential, must agree to use adequate contraception starting with the first dose of study medication through 120 days after the last dose of study medication or through 180 days after last dose of chemotherapeutic agents.

Exclusion Criteria:

* Has predominantly squamous cell histology NSCLC.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks prior to administration of pembrolizumab.
* Before the first dose of study medication: a) Has received prior systemic cytotoxic chemotherapy for metastatic disease, b) Has received antineoplastic biological therapy (e.g., erlotinib, crizotinib, cetuximab), c) Had major surgery (<3 weeks prior to first dose)
* Received radiation therapy to the lung that is >30 Gray (Gy) within 6 months of the first dose of study medication.
* Completed palliative radiotherapy within 7 days of the first dose of study medication.
* Is expected to require any other form of antineoplastic therapy while on study.
* Received a live-virus vaccination within 30 days of planned start of study medication.
* Has clinically active diverticulitis, intra-abdominal abscess, gastrointestinal obstruction, peritoneal carcinomatosis.
* Known history of prior malignancy except if participant has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy, except for successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, or other in situ cancers.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Previously had a severe hypersensitivity reaction to treatment with another monoclonal antibody (mAb).
* Known sensitivity to any component of cisplatin, carboplatin or pemetrexed.
* Has active autoimmune disease that has required systemic treatment in past 2 years.
* Is on chronic systemic steroids.
* Is unable to interrupt aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs), other than an aspirin dose ≤1.3 g per day, for a 5-day period (8-day period for long-acting agents, such as piroxicam).
* Is unable or unwilling to take folic acid or vitamin B12 supplementation.
* Had prior treatment with any other anti-programmed cell death-1 (PD-1), or PD-ligand 1 (PD-L1) or PD-L2 agent or an antibody targeting other immuno-regulatory receptors or mechanisms. Has participated in any other pembrolizumab study and has been treated with pembrolizumab.
* Has an active infection requiring therapy.
* Has known history of Human Immunodeficiency Virus (HIV).
* Has known active Hepatitis B or C.
* Has known psychiatric or substance abuse disorder that would interfere with cooperation with the requirements of the trial.
* Is a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of substance abuse (including alcohol).
* Has symptomatic ascites or pleural effusion.
* Has interstitial lung disease or a history of pneumonitis that required oral of IV glucocorticoids to assist with management.
* Is pregnant or breastfeeding, or expecting to conceive or father children prior to 120 days after the last dose of study medication or through 180 days after last dose of chemotherapeutic agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2023-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Garassino MC, Cheng Y, Rodriguez-Abreu D, Novello S, Mazieres J, Robinson AG, Powell SF, Halmos B, Gray JE, Wang M, Chen C, Yang J, Souza F, Schwarzenberger P, Paz-Ares L. Impact of Tumor Response and Response Duration on Survival Among Participants Receiving Pembrolizumab Plus Chemotherapy as First-Line Therapy for Non-Small-Cell Lung Cancer. Oncol Ther. 2025 Sep;13(3):667-681. doi: 10.1007/s40487-025-00350-6. Epub 2025 Jun 11. PMID 40498298
- [Derived] Cheng Y, Yang JC, Okamoto I, Zhang L, Hu J, Wang D, Hu C, Zhou J, Wu L, Cao L, Liu J, Zhang H, Sun H, Wang Z, Gao H, Yan Y, Xiao S, Lin J, Pietanza MC, Kurata T. Pembrolizumab plus chemotherapy for advanced non-small-cell lung cancer without tumor PD-L1 expression in Asia. Immunotherapy. 2023 Sep;15(13):1029-1044. doi: 10.2217/imt-2023-0043. Epub 2023 Jul 19. PMID 37465924
- [Derived] Garassino MC, Gadgeel S, Speranza G, Felip E, Esteban E, Domine M, Hochmair MJ, Powell SF, Bischoff HG, Peled N, Grossi F, Jennens RR, Reck M, Hui R, Garon EB, Kurata T, Gray JE, Schwarzenberger P, Jensen E, Pietanza MC, Rodriguez-Abreu D. Pembrolizumab Plus Pemetrexed and Platinum in Nonsquamous Non-Small-Cell Lung Cancer: 5-Year Outcomes From the Phase 3 KEYNOTE-189 Study. J Clin Oncol. 2023 Apr 10;41(11):1992-1998. doi: 10.1200/JCO.22.01989. Epub 2023 Feb 21. PMID 36809080
- [Derived] Garassino MC, Gadgeel S, Novello S, Halmos B, Felip E, Speranza G, Hui R, Garon EB, Horinouchi H, Sugawara S, Rodriguez-Abreu D, Reck M, Cristescu R, Aurora-Garg D, Loboda A, Lunceford J, Kobie J, Ayers M, Piperdi B, Pietanza MC, Paz-Ares L. Associations of Tissue Tumor Mutational Burden and Mutational Status With Clinical Outcomes With Pembrolizumab Plus Chemotherapy Versus Chemotherapy For Metastatic NSCLC. JTO Clin Res Rep. 2022 Nov 8;4(1):100431. doi: 10.1016/j.jtocrr.2022.100431. eCollection 2023 Jan. PMID 36793385
- [Derived] Garon EB, Aerts J, Kim JS, Muehlenbein CE, Peterson P, Rizzo MT, Gadgeel SM. Safety of pemetrexed plus platinum in combination with pembrolizumab for metastatic nonsquamous non-small cell lung cancer: A post hoc analysis of KEYNOTE-189. Lung Cancer. 2021 May;155:53-60. doi: 10.1016/j.lungcan.2021.02.021. Epub 2021 Feb 19. PMID 33730652
- [Derived] Gadgeel S, Rodriguez-Abreu D, Speranza G, Esteban E, Felip E, Domine M, Hui R, Hochmair MJ, Clingan P, Powell SF, Cheng SY, Bischoff HG, Peled N, Grossi F, Jennens RR, Reck M, Garon EB, Novello S, Rubio-Viqueira B, Boyer M, Kurata T, Gray JE, Yang J, Bas T, Pietanza MC, Garassino MC. Updated Analysis From KEYNOTE-189: Pembrolizumab or Placebo Plus Pemetrexed and Platinum for Previously Untreated Metastatic Nonsquamous Non-Small-Cell Lung Cancer. J Clin Oncol. 2020 May 10;38(14):1505-1517. doi: 10.1200/JCO.19.03136. Epub 2020 Mar 9. PMID 32150489
- [Derived] Garassino MC, Gadgeel S, Esteban E, Felip E, Speranza G, Domine M, Hochmair MJ, Powell S, Cheng SY, Bischoff HG, Peled N, Reck M, Hui R, Garon EB, Boyer M, Wei Z, Burke T, Pietanza MC, Rodriguez-Abreu D. Patient-reported outcomes following pembrolizumab or placebo plus pemetrexed and platinum in patients with previously untreated, metastatic, non-squamous non-small-cell lung cancer (KEYNOTE-189): a multicentre, double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2020 Mar;21(3):387-397. doi: 10.1016/S1470-2045(19)30801-0. Epub 2020 Feb 6. PMID 32035514
- [Derived] Gandhi L, Rodriguez-Abreu D, Gadgeel S, Esteban E, Felip E, De Angelis F, Domine M, Clingan P, Hochmair MJ, Powell SF, Cheng SY, Bischoff HG, Peled N, Grossi F, Jennens RR, Reck M, Hui R, Garon EB, Boyer M, Rubio-Viqueira B, Novello S, Kurata T, Gray JE, Vida J, Wei Z, Yang J, Raftopoulos H, Pietanza MC, Garassino MC; KEYNOTE-189 Investigators. Pembrolizumab plus Chemotherapy in Metastatic Non-Small-Cell Lung Cancer. N Engl J Med. 2018 May 31;378(22):2078-2092. doi: 10.1056/NEJMoa1801005. Epub 2018 Apr 16. PMID 29658856
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26082&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eighty-four participants randomized to receive Control switched over to receive pembrolizumab monotherapy. Participants receiving pembrolizumab in first course and those switching over from placebo to pembrolizumab monotherapy were eligible to receive second course of pembrolizumab monotherapy if they met certain criteria. Data from second course treatment contributed to safety data only. All primary and secondary outcome measures are based on protocol-specified cutoff (2017-11-08).
Groups:
- Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed: Participants received pembrolizumab 200 mg IV PLUS pemetrexed 500 mg/m^2 IV (with vitamin supplementation) PLUS cisplatin 75 mg/m^2 IV OR carboplatin AUC 5 IV on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by pembrolizumab 200 mg IV PLUS pemetrexed 500 mg/m^2 IV Q3W until progression. (Participants who received pembrolizumab 200 mg IV Q3W for up to 2 years but experienced disease progression, were eligible to receive a second course of pembrolizumab monotherapy 200 mg IV Q3W, at the investigator's discretion, for up to 1 additional year.)
- Control: Participants received saline placebo IV PLUS pemetrexed 500 mg/m^2 IV (with vitamin supplementation) PLUS cisplatin 75 mg/m^2 IV OR carboplatin AUC 5 IV on Day 1 of every 3-week cycle (Q3W) for 4 cycles followed by saline placebo IV PLUS pemetrexed 500 mg/m^2 IV Q3W until progression. (Effective 23-Dec-2019, participants discontinued saline placebo. If documented disease progression had occurred, and participants receiving Control met certain criteria, they were eligible to switch over to receive pembrolizumab monotherapy Q3W for the remainder of the study.)
Period: Overall Study
Arm/Group | Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed | Control
Started | 410 | 206
Treated | 405 | 202
Switched to Pembrolizumab | 0 | 84
Completed | 0 | 0
Not Completed | 410 | 206
Not completed — Death | 329 | 181
Not completed — Lost to Follow-up | 3 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Sponsor Decision | 64 | 13
Not completed — Withdrawal by Subject | 13 | 9

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population consisted of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed | Control | Total
Number analyzed (Participants) | 410 | 206 | 616
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (9.4) | 62.8 (9.1) | 63.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 156 | 97 | 253
  Male | 254 | 109 | 363
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 10 | 8 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 3 | 14
  White | 387 | 195 | 582
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Programmed Cell Death-Ligand 1 (PD-L1) Tumor Status [Count of Participants; unit: Participants] — Participants were assessed for their PD-L1 tumor expression level by immunohistochemistry assay using tumor tissue from an archival or newly obtained biopsy. Participants with a TPS ≥1% were classified as PD-L1 positive and participants with a TPS <1% were classified as PD-L1 negative.
  Participants
    TPS <1% | 127 | 63 | 190
    TPS ≥1% | 260 | 128 | 388
    Not Evaluable | 23 | 15 | 38
Platinum Chemotherapy [Count of Participants; unit: Participants] — Participants were classified according to the type of platinum chemotherapy the Investigator chose for them to receive: Cisplatin or Carboplatin.
  Participants
    Cisplatin | 113 | 58 | 171
    Carboplatin | 297 | 148 | 445
Smoking Status [Count of Participants; unit: Participants] — Participants were classified according to their smoking status: Never Smoker or Former/Current Smoker.
  Participants
    Never Smoker | 48 | 25 | 73
    Former/Current Smoker | 362 | 181 | 543

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as Assessed by Blinded Central Imaging
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. The PFS per RECIST 1.1 is presented.
Time Frame: Up to approximately 21 months
Population: The analysis population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed | Control
Number analyzed (Participants) | 410 | 206
Months | 8.8 [7.6 to 9.2] | 4.9 [4.7 to 5.5]
Statistical Analysis 1: Comparison: Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed vs Control; Test type: Superiority; p < 0.00001, Log Rank; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.43 to 0.64] — Based on Cox regression model with treatment as a covariate stratified by PD-L1 status (≥1% vs. <1%), platinum chemotherapy (cisplatin vs. carboplatin) & smoking status (never vs. former/current). Pembrolizumab=numerator; Control=denominator

2. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the interim analysis were censored at the date of the last follow-up. The OS is presented.
Time Frame: Up to approximately 21 months
Population: The analysis population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed | Control
Number analyzed (Participants) | 410 | 206
Months | NA [NA to NA] — NA=Median OS not reached NA=Lower Limit OS not reached NA=Upper Limit OS not reached | 11.3 [8.7 to 15.1]
Statistical Analysis 1: Comparison: Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed vs Control; Test type: Superiority; p < 0.00001, Log Rank; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.38 to 0.64] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Overall Response Rate (ORR) Per RECIST 1.1 as Assessed by Blinded Central Imaging
Description: ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1. The percentage of participants who experienced a CR or PR is presented.
Time Frame: Up to approximately 21 months
Population: The analysis population consisted of all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed | Control
Number analyzed (Participants) | 410 | 206
Percentage of Participants | 47.6 [42.6 to 52.5] | 18.9 [13.8 to 25.0]
Statistical Analysis 1: Comparison: Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed vs Control; Test type: Superiority; p < 0.0001, Stratified Miettinen and Nurminen — H0:Difference in percentages=0 vs H1:Difference in percentages>0; Difference in Percentage vs. Control = 28.5, 95% CI 2-sided [21.1 to 35.4] — Miettinen and Nurminen method with treatment as a covariate stratified by PD-L1 status (≥1% vs. <1%), platinum chemotherapy (cisplatin vs. carboplatin) & smoking status (never vs. former/current). Pembrolizumab=numerator; Control=denominator

4. Secondary Outcome: Duration of Response (DOR) Per RECIST 1.1 as Assessed by Blinded Central Imaging
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR was defined as the time from first documented evidence of a CR or PR until PD or death. DOR for participants who had not progressed or died at the time of analysis was to be censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. DOR assessments were based on blinded central imaging review with confirmation. The DOR per RECIST 1.1 for all participants who experienced a confirmed CR or PR is presented.
Time Frame: Up to approximately 21 months
Population: The analysis population consisted of all randomized participants who experienced a confirmed CR or confirmed PR.
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed | Control
Number analyzed (Participants) | 195 | 39
Months | 11.2 [1.1 to 18.0] | 7.8 [2.1 to 16.4]

5. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a study participant administered study drug and which does not necessarily have to have a causal relationship with this study drug. The number of participants who experienced an AE is presented.
Time Frame: Up to approximately 21 months (Serious AEs: Up to 90 days after last dose of study treatment; Other AEs: Up to 30 days after last dose of study treatment)
Population: The analysis population consisted of all randomized participants who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed | Control
Number analyzed (Participants) | 405 | 202
Participants | 404 | 200

6. Secondary Outcome: Number of Participants Who Discontinued Any Study Drug Due to an AE
Description: An AE was defined as any untoward medical occurrence in a study participant administered study drug and which does not necessarily have to have a causal relationship with this study drug. The number of participants who discontinued any randomized study drug due to an AE is presented.
Time Frame: Up to approximately 21 months
Population: The analysis population consisted of all randomized participants who received ≥1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed | Control
Number analyzed (Participants) | 405 | 202
Participants | 112 | 30

7. Other Pre Specified Outcome: Progression-Free Survival (PFS) as Assessed by Investigator Immune-related RECIST (irRECIST) Response Criteria
Description: PFS was defined as the time from randomization to the first documented immune-related progressive disease (irPD) or death due to any cause, whichever occurred first. Per irRECIST, irPD was confirmed if any of the following are observed in 2 scans performed at least 4 weeks apart: target lesion sum of diameters remains ≥20 % and at least 5 mm absolute increase compared to nadir; non-target disease resulting in initial PD is qualitatively worse; new lesion resulting in initial irPD is qualitatively worse; additional new lesion(s) since last evaluation; or additional new non-target lesion progression since last evaluation. The PFS per irRECIST 1.1 is presented.
Time Frame: Up to approximately 39 months
Population: The analysis population consisted of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed | Control
Number analyzed (Participants) | 410 | 206
Months | 10.3 [9.0 to 11.3] | 5.0 [4.8 to 6.0]
Statistical Analysis 1: Comparison: Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed vs Control; Test type: Superiority; p < 0.00001, Log Rank; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.41 to 0.59] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to approximately 88 months
Description: Safety Population: All participants receiving ≥1 dose of randomized study drug. All-Cause Mortality Population: All randomized participants. Per protocol, progression of cancer under study was not considered an AE unless related to study drug. Therefore, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" & "Disease progression" not related to study drug are excluded as AEs.
Groups:
- Control Switched Over to Pembrolizumab Monotherapy: Qualified participants who received saline placebo with pemetrexed and platinum chemotherapy followed by placebo and pemetrexed, and who experienced disease progression, were switched over to receive pembrolizumab monotherapy 200 mg IV on Day 1 Q3W for up to 2 years.
- Control Switched Over to Pembrolizumab Monotherapy (Second Course): Participants who were switched from saline placebo to receive pembrolizumab monotherapy, and met certain criteria, received a second course of pembrolizumab monotherapy at 200 mg IV Q3W for up to 1 additional year.
- Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed (Second Course): Participants who received pembrolizumab PLUS pemetrexed and platinum chemotherapy followed by pembrolizumab PLUS pemetrexed during the initial treatment but experienced disease progression, and met certain criteria, received a second course of pembrolizumab monotherapy at 200 mg IV Q3W for up to 1 additional year.
Arm/Group | Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed | Control | Control Switched Over to Pembrolizumab Monotherapy | Control Switched Over to Pembrolizumab Monotherapy (Second Course) | Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed (Second Course)
All-Cause Mortality (participants affected / at risk) | 330/410 | 113/206 | 74/84 | 1/2 | 4/9
Serious Adverse Events (participants affected / at risk) | 233/405 | 102/202 | 29/84 | 0/2 | 2/9
Other Adverse Events (participants affected / at risk) | 395/405 | 196/202 | 64/84 | 2/2 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed (N=405) | Control (N=202) | Control Switched Over to Pembrolizumab Monotherapy (N=84) | Control Switched Over to Pembrolizumab Monotherapy (Second Course) (N=2) | Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed (Second Course) (N=9)
Anaemia (Blood and lymphatic system disorders) | 13 (14) | 11 (12) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 25 (26) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 11 (11) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 13 (14) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myopericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 14 (16) | 5 (8) | 0 (0) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip oedema (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mesenteric artery embolism (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 7 (8) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Asthenia (General disorders) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 6 (6) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 9 (10) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis sclerosing (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacillus bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
CNS ventriculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 5 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 34 (35) | 18 (21) | 4 (4) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Salmonella bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 7 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tuberculous pleurisy (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 2 (5) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shoulder fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 5 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertrophic osteoarthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Central nervous system vasculitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Demyelinating polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacunar stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 11 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 4 (5) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 5 (6) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4) | 3 (4) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin sensitisation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed (N=405) | Control (N=202) | Control Switched Over to Pembrolizumab Monotherapy (N=84) | Control Switched Over to Pembrolizumab Monotherapy (Second Course) (N=2) | Pembrolizumab+Pemetrexed+Platinum Chemotherapy Followed by Pembrolizumab+Pemetrexed (Second Course) (N=9)
Anaemia (Blood and lymphatic system disorders) | 186 (253) | 91 (114) | 6 (8) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 26 (44) | 13 (18) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 108 (213) | 49 (92) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 68 (108) | 25 (37) | 1 (1) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 14 (19) | 11 (12) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 17 (21) | 4 (7) | 1 (2) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 31 (38) | 5 (7) | 6 (6) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 21 (23) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 75 (87) | 22 (24) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 39 (49) | 13 (14) | 7 (7) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 29 (31) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 143 (220) | 67 (87) | 7 (7) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 123 (179) | 41 (54) | 11 (19) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 28 (31) | 11 (11) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 17 (18) | 6 (6) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 232 (430) | 103 (186) | 16 (18) | 0 (0) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 37 (54) | 16 (21) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 104 (183) | 43 (70) | 12 (14) | 0 (0) | 1 (2)
Asthenia (General disorders) | 85 (158) | 47 (74) | 6 (8) | 0 (0) | 0 (0)
Chest pain (General disorders) | 38 (44) | 12 (14) | 6 (6) | 0 (0) | 0 (0)
Fatigue (General disorders) | 173 (285) | 80 (127) | 8 (9) | 0 (0) | 1 (1)
Mucosal inflammation (General disorders) | 37 (48) | 16 (24) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 103 (180) | 35 (48) | 11 (11) | 0 (0) | 0 (0)
Pain (General disorders) | 22 (22) | 7 (7) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 84 (118) | 30 (47) | 6 (7) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 23 (29) | 6 (7) | 2 (2) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 37 (48) | 18 (33) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 11 (12) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 47 (76) | 10 (12) | 5 (6) | 0 (0) | 2 (2)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 21 (29) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 10 (12) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 44 (59) | 16 (17) | 1 (1) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 34 (47) | 13 (17) | 4 (6) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 50 (63) | 19 (23) | 4 (4) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 40 (57) | 13 (16) | 5 (6) | 1 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 16 (21) | 9 (11) | 2 (2) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 58 (97) | 17 (29) | 4 (10) | 1 (1) | 0 (0)
Blood magnesium decreased (Investigations) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Tri-iodothyronine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 44 (59) | 16 (17) | 4 (4) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 28 (57) | 13 (20) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 122 (172) | 63 (81) | 17 (19) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 34 (49) | 7 (10) | 2 (2) | 1 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 51 (91) | 16 (20) | 2 (2) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 37 (54) | 8 (14) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 24 (38) | 5 (13) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 70 (99) | 28 (33) | 10 (12) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 71 (86) | 26 (29) | 7 (7) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 19 (23) | 7 (7) | 2 (2) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10 (13) | 8 (9) | 1 (1) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 16 (16) | 6 (8) | 4 (4) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 37 (47) | 18 (18) | 6 (7) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 58 (64) | 22 (27) | 2 (2) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 36 (41) | 17 (17) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 57 (72) | 22 (29) | 5 (7) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 24 (33) | 14 (21) | 1 (1) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 31 (35) | 17 (17) | 1 (1) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 104 (139) | 62 (71) | 9 (13) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 97 (118) | 51 (59) | 15 (20) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 29 (35) | 7 (11) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 16 (20) | 2 (2) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 27 (33) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 27 (33) | 9 (10) | 3 (4) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 25 (28) | 10 (10) | 1 (1) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 22 (24) | 10 (10) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 27 (28) | 20 (22) | 1 (1) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 30 (38) | 4 (5) | 3 (3) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 59 (80) | 23 (25) | 4 (4) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 89 (131) | 27 (36) | 4 (4) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 23 (25) | 11 (14) | 5 (6) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 24 (27) | 4 (4) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/80/NCT02578680/Prot_SAP_001.pdf